CLINICAL TRIAL: NCT00860223
Title: An Open-Label, Nonrandomized, Crossover Study to Evaluate the Potential Effect of Multiple Doses of Neratinib on the Pharmacokinetics of a Single Dose of Digoxin When Administered Orally to Healthy Adult Subjects
Brief Title: Study Evaluating The Potential Effect Of Multiple Doses Of Neratinib On The Pharmacokinetics Of A Single Dose Of Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-1119
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Digoxin; neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Digoxin alone
  Interventions: Drug: Digoxin
- 2 (Experimental): Digoxin plus neratinib
  Interventions: Drug: Digoxin; Drug: Neratinib

INTERVENTIONS:
Drug: Digoxin
Drug: Neratinib — HKI-272
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the potential effect of multiple doses of neratinib on the pharmacokinetics (how the body absorbs, distributes, metabolizes and/or excretes) of a single dose of digoxin.

ELIGIBILITY:
Inclusion criteria:

* Healthy men and women of non-childbearing potential, age 18-50

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: concentration of digoxin in blood and urine | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Miami, Florida, United States